CLINICAL TRIAL: NCT06508697
Title: CT-Angiography-Derived Plaque Characteristics on Cardiac Events in Deferral Patients by Invasive Fractional Flow Reserve
Brief Title: CT-Angiography Plaque Characteristics and Events in Deferral Patients by Invasive Fractional Flow Reserve
Acronym: CAPTURE
Status: Recruiting | Type: Observational
Sponsor: Fujita Health University (Other)
Responsible Party: Principal Investigator, Yukio Ozaki, Professor of Cardiology, Fujita Health University
Other Study IDs: CI20-015
Record Dates: First submitted 2024-07-14; First posted 2024-07-18 (Actual); Last update posted 2025-01-03 (Actual); Status verified 2024-07

CONDITIONS: Patient Preference
MeSH Terms: conditions — Patient Preference

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients who underwent CTA within 90 days before ICA with FFR pressure: A consecutive series of patients who underwent Coronary computed tomography angiography (CTA) within 90 days before invasive coronary angiography (ICA) with fractional flow reserve (FFR) pressure measurement were candidates for this study at Fujita Health University Hospital, Bantane Hospital, and Nagoya First Red Cross Hospital.
  Interventions: Diagnostic Test: invasive coronary angiography (ICA) with fractional flow reserve (FFR) pressure measurement

INTERVENTIONS:
Diagnostic Test: invasive coronary angiography (ICA) with fractional flow reserve (FFR) pressure measurement — A consecutive series of patients who underwent Coronary computed tomography angiography (CTA) within 90 days before invasive coronary angiography (ICA) with fractional flow reserve (FFR) pressure measurement were candidates for this study at Fujita Health University Hospital, Bantane Hospital, and Nagoya First Red Cross Hospital
  Other Names: Coronary computed tomography angiography (CTA)

SUMMARY:
Fractional flow reserve (FFR)-guided PCI for chronic coronary syndromes (CCS) is reported to improve the outcomes compared with angiography-guided PCI. However, cardiac-events still occur in FFR-deferral patients in long-term follow-up. Coronary computed tomography angiography (CTA)-defined high-risk-plaque (HRP) is known to relate future cardiac events. The investigators hypothesized that CTA might identify plaque features linked to future cardiac events in deferral patients.

DETAILED DESCRIPTION:
Although fractional flow reserve (FFR)-guided percutaneous-coronary-intervention (PCI) has improved short- and middle-term outcome compared with angiography-guided PCI alone, cardiac-events still occur in FFR-deferral patients in long-term.1-4 Recent J-CONFIRM registry examined 1263 patients with 1447 lesions in whom revascularization was deferred based on FFR in the 28 centers.5 While 2-year target vessel failure (TVF) rate was 5.5% in deferred lesions in the J-CONFIRM registry, 5-year TVF raised up 11.6% in deferred lesions.5, 6 The TVF rate raised up from 5.5% to 11.6% in the last 3 years mainly due to clinically driven target-vessel-revascularization (TVR) in the registry.5, 6 In the DEFER trial, patients with FFR > 0.75 were randomly assigned to PCI deferral (Defer) or performance (Perform) and patients showing FFR < 0.75 underwent PCI (Reference).3 The 5-year cardiac death and acute myocardial infarction (AMI) rate were excellent in the Defer group as compared to Perform and Reference groups (3.3%, 7.9%, and 15.7%, p < 0.003, respectively).4 However, 15-year follow-up of the DEFER study revealed that all cause of mortality and TVR were similar among Defer, Perform and Reference groups (mortality; 33.0% vs. 31.1% vs. 36.1% p= 0.441 respectively, and TVR; 36.3% vs. 27.8% vs. 35.4%, p= 0.522 respectively).7 Favorable initial 5-year clinical outcome in deferral patients has been lost during 15-year follow-up in the DEFER study. It is urgent issue to disclose the factor to predict future cardiac events in deferral lesions. The failure of PCI to modify long-term outcomes may stem from its inability to modify the underlying atherosclerotic process.

Furthermore, recent PREVENT study disclosed that in patients with non-flow-limiting (FFR >0.80) vulnerable coronary plaques identified by intracoronary imaging, preventive PCI reduced major adverse cardiac events (MACE) arising from high-risk vulnerable plaques, compared with optimal medical therapy (OMT) alone8. Although their high-risk vulnerable plaques were defined using intracoronary imaging but not coronary CT angiography (CTA) in the PREVENT study, the presence of high-risk vulnerable plaque without flow-limiting (FFR >0.80) frequently caused the subsequent cardiac events in patients without the initial PCI.

While CTA is known to be useful to evaluate coronary artery plaque features as well as stenosis severity, high-risk plaque (HRP) on coronary CTA defined as a combination of positive remodeling (PR) and low attenuation plaque (LAP) has been reported to be associated with the future cardiac events.9-12 Gallone and coworkers reported in their meta-analysis that high-risk coronary plaque characteristics significantly predicted patient-level and lesion-level major adverse cardiac event (MACE) in the future, using various high-risk coronary plaque definitions by several intracoronary imaging modalities and CTA.13 The investigators hypothesized that CTA could identify plaque features linked to future cardiac events in deferral patients. To determine the predictive factors for future cardiac events in FFR-based deferral patients, the investigators examined clinical features and plaque characteristics on CTA in the deferral lesions based on invasive FFR in consecutive 373 patients with chronic coronary syndromes (CCS).

ELIGIBILITY:
Inclusion Criteria:

* men and women aged ≥20 years,
* patients having chronic coronary syndromes (CCS,
* Coronary computed tomography angiography (CTA) was performed within 90 days before invasive coronary angiography (ICA) with fractional flow reserve (FFR) pressure measurement.

Exclusion Criteria:

* patients with a history of coronary bypass grafting (CABG) because CABG changed local coronary flow dynamics,
* patients with left-main disease,
* patients with fractional flow reserve (FFR) in stented vessels due to inability to estimate plaque morphology in the stented lesion by coronary computed tomography angiography.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: A consecutive series of 437 patients who underwent CTA within 90 days before ICA with FFR pressure measurement were candidates for this study at Fujita Health University Hospital, Bantane Hospital, and Nagoya First Red Cross Hospital
Sampling Method: Non-Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2025-01-30 (Estimated); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Cardiac events in patient level | From 2018 to 2026
  a composite of cardiac death, non-fatal acute coronary syndrome (ACS), and ischemia-driven revascularization for patient-level analysis
Cardiac events in lesion level | From 2018 to 2026
  lesion-level ACS and lesion-level ischemia-driven revascularization

CONTACTS AND LOCATIONS:
Overall Officials: YUKIO OZAKI, MD, PhD, Principal Investigator — Fujita Health University, Aichi, Japan
Locations (1):
- Fujita Health University, Toyoake, Aichi-ken, Japan